CLINICAL TRIAL: NCT01698216
Title: Switching From Risperidone Long Acting Injection (Consta®) to Paliperidone Palmitate (Sustenna®) in Patients With Schizophrenia and Its Influence on Subjective Well-Being: A Prospective Observational Study
Brief Title: Switching From Consta® to Sustenna® in Patients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yong Min Ahn, professor, Seoul National University Hospital
Other Study IDs: Consta_Sustenna
Record Dates: First submitted 2012-09-27; First posted 2012-10-02 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Schizophrenia
Keywords: Paliperidone; Palmitate; switching; schizophrenia; subjective well-being
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Consta Sustenna switching: The patients group who switched to paliperidone palmitate from risperidone long acting injection

SUMMARY:
The aim of this study is observation of effectiveness and side effect of patients with schizophrenia who will switch the antipsychotics from risperidone long acting injection to paliperidone palmitate.

DETAILED DESCRIPTION:
In this study, investigators are going to enroll the patients who will switch the risperidone long acting injection to paliperidone palmitate. And investigators will examine the effectiveness and side effect of paliperidone palmitate. In addition, effectiveness and side effect related variables will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 ~ 65
* Patient with schizophrenia according to DSM-IV criteria
* Patient have signed on the informed consent, and well understood the objective and procedure of this study.
* Maintenance therapy more than 6 months with Risperidone Long Acting Injection monotherapy or other with concomitant antipsychotics, and stable dose of Risperidone Long Acting Injection was maintained 8 weeks more. The stable dose of other antipsychotics has been maintained 8 months and more.
* Patient wants to switch antipsychotics to Paliperidone Palmitate.
* PANSS total score ≤ 80
* Each score of conceptual disorganization(P2), hallucinatory behavior(P3), Suspiciousness/persecution(P6), unusual thought content(G9)in PANSS ≤ 4
* Competent patient who is manage to answer the questionnaires.
* In case of female at child-bearing age, consent to use appropriate contraceptive methods(oral pill, contraceptive injection, intrauterine device, double barrier method and contraceptive patch) during entire duration of this study.

Exclusion Criteria:

* No history of antipsychotics use.
* Past history of NMS.
* Allergy or hypersensitivity to Risperidone or Paliperidone ER.
* Concomitant antipsychotics was oral Risperidone or Paliperidone ER.
* Initiating or dose-changing of SSRI, MAOI, TCA within 2 months(maintenance is allowed if those have been stable for at least 30days prior to study entry and would not be any dose changes during the study)
* Initiating of Lithium, Valproic acid, Carbamazepine, Topiramate, Lamotrigine or other mood stabilizer within 2months (maintenance is allowed).
* Patient who is supposed to be impossible to participate to this study due to clinical risk of suicide or aggressive behavior based on clinician's opinion.
* Current substance dependence(DSM-IV) or past history of dependence (more than 6months)
* Significant biochemical or hematological abnormality or abnormal finding of urinalysis, based on clinician's opinion.
* History of cardiac disease which predispose to QT prolongation(sick sinus, complete AV block, CHF, ventricular tachycardia, hypokalemia or hypocalcemia) or current medication of QT prolonging drugs
* Pregnant or breast-feeding female patient.
* History of participating to other investigational drug trial within 1month prior to screening.
* Investigator or employee at clinical trial center, personnel related to investigator or trial center on this or other study, or family of employee or investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with schizophrenia who would be switched to Paliperidone Palmitate from Risperidone Long Acting Injection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Subjective Well-being Under Neuroleptic Treatment (SWN) | Change from Baseline in SWN score at 108 weeks

SECONDARY OUTCOMES:
Korean Drug Attitude Inventory-10 | Change from Baseline in score at 108 weeks
Positive and Negative Syndrome Scale | 0,4,8,16,24,36,48,60,72,84,96,108 week
Clinical Global Impression-Severity, Improvement | 0,4,8,16,24,36,48,60,72,84,96,108 week
Personal and Social Performance Scale | 0,4,8,16,24,36,48,60,72,84,96,108 week
Symptom Check List-90-Revised | 0,4,8,16,24,36,48,60,72,84,96,108 week
Drug-Induced ExtraPyramidal Symptoms Scale | 0,4,8,16,24,36,48,60,72,84,96,108 week
Liverpool University Neuroleptic Side Effect Rating Scale | 0,4,8,16,24,36,48,60,72,84,96,108 week
Visual Analog Scale | 0,4,8,16,24,36,48,60,72,84,96,108 week
  injection site pain
ECG | 8, 24, 48, 72, 108 week
  electrocardiogram
blood pressure | 0,4,8,16,24,48,72,108 week
Body weight | 0,4,8,16,24,48,72,108 week
waist circumference | 0,4,8,16,24,48,72,108 week

CONTACTS AND LOCATIONS:
Overall Officials: Yong Min Ahn, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea